CLINICAL TRIAL: NCT04233229
Title: Evaluation of a Closed-loop Insulin Delivery System at Home With Tailored Home Care Services in Poorly Controlled Type 2 Diabetes: a Randomized Controlled Trial vs Usual Care
Brief Title: Evaluation of a Closed-loop Insulin Delivery System at Home With Tailored Home Care Services in Poorly Controlled Type 2 Diabetes Patients (T2D)
Acronym: CLOSEAP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALMED-19-003
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- closed-loop and home care services (Experimental): automated insulin delivery system (Closed-loop) with tailored Home Healthcare Provider (HHP) services
  Interventions: Device: t:slim X2 with Control-IQ; Other: home healthcare services
- usual care (Active Comparator): multiple daily injection insulin regimen with family nurse's daily assistance at home for performing insulin injections and/or glucose monitoring
  Interventions: Other: usual care for daily insulin treatment

INTERVENTIONS:
Device: t:slim X2 with Control-IQ — closed-loop in patients at home for three months
  Arms: closed-loop and home care services
Other: home healthcare services — home healthcare services from Air Liquide in patients at home for three months
  Arms: closed-loop and home care services
Other: usual care for daily insulin treatment — multiple daily injection insulin regimen with family nurse's daily assistance at home for performing insulin injections and/or glucose monitoring
  Arms: usual care

SUMMARY:
Closed-loop insulin delivery system has the potential to improve the condition of many poorly controlled insulin-treated Type 2 Diabetes (T2D) patients.

A wide acceptance of the Artificial Pancreas (AP) usage in T2D care will strongly depend on the identification of subpopulations and care settings where the AP could significantly improve the risk- and cost-benefit balances of T2D management as compared to established practice.

The aim of this interventional study, therefore, is to investigate whether a therapeutic solution combining an automated insulin delivery AP system with a tailored Home Healthcare Provider (HHP) service can improve blood glucose control, reduce the rate of acute metabolic complications (hypoglycaemia and hyperglycaemia), improve both the patients quality of life and experience, and reduce the healthcare related costs in patients with uncontrolled T2D needing home nursing care for their daily insulin treatment versus usual care.

ELIGIBILITY:
Selection criteria:

* 1. Male or female patient aged 18 years or older, 2. Type 2 Diabetes diagnosed for at least 6 months with a stable authorized antidiabetic therapeutic regimen for 3 months, 3. Treated with insulin for at least 6 months, 4. Patient with 8.0% ≤ HbA1c <12.0% within the last 3 months before selection, 5. Patient with a current minimum of 2 daily insulin injections and who would benefit of an optimisation, 6. Patient requiring long term family nurse's daily assistance at home for performing insulin injections and/or glucose monitoring, 7. Total daily insulin dose < 1.5 U/kg, 8. Patient willing and able to complete the requirements of the study, 9.Patient living with a caregiver or a diabetes care partner, or patient living alone but with a caregiver living nearby who has a telephone and a key to his or her home, 10.Patient living in an area covered by a GSM (Global System for Mobile Communications) network and not considering a trip outside of France or out of an area covered by a GSM network within the planned dates corresponding to the 30 days of the installation of the pump (to cover the open-loop period and first 15 days of the closed-loop period), and the last 20 days of the study.

Inclusion Criteria:

1. Patient having demonstrated ability to understand the benefits and harms of the automated insulin delivery system and to continuously and safely wear a CGM (Continuous Glucose Monitor), as per investigator's judgement,
2. Family nurse having demonstrated ability to use the automated insulin delivery system, as per HHP judgement,
3. Patient able to use basic technology such as a cell phone and having demonstrated ability to use the automated insulin delivery system, as per Home Healthcare Provider (HHP) judgment. In case the patient has not demonstrated ability to use the automated insulin delivery system, his (her) caregiver has to demonstrate ability to use basic technology such as a cell phone and the automated insulin delivery system instead as per Home Healthcare Provider (HHP) judgment. The caregiver has to be an adult person able to speak and read French, having demonstrated ability to use the automated insulin delivery system, with no known medical condition that in the judgment of the investigator might interfere with the completion of the protocol. The caregiver must have committed to maintain uninterrupted availability via personal cell phone and to provide assistance to the patient and must be knowledgeable at all times of the participant's location during the day when closed loop is in use.
4. 14 days completed (ie ≥ 70% of the daily data points non missing) CGM data from the selection period (the CGM period may be repeated only once if uncompleted data),
5. Patient covered by healthcare insurance (in accordance with French regulation),
6. Patient who has received verbal and written information about the study and who signed the informed consent form before any study related procedure.
7. Patient under curatorship must have received the agreement of their legal guardian to participate to the study.

Exclusion Criteria:

1. Pregnant or breastfeeding woman,
2. Patient who experienced a severe hypoglycaemic event having led to a hospitalisation or having required a third party assistance within the past 6 months,
3. Patient who experienced a diabetic ketoacidosis within the past 6 months,
4. Patient who has demonstrated a marked decrease in hypoglycaemia perception defined by a Gold score > 4,
5. Patient who has disabilities which could compromise the compliance to the study, in the investigator's opinion,
6. Patient with severe health impairment resulting in short life expectancy (< 1 year) as assessed by the investigator,
7. Patient participating in another interventional or observational clinical trial or who participated in another interventional clinical trial within 30 days before selection,
8. Patient known allergy to any component of the automated insulin delivery system compounds,
9. Proliferative retinopathy (assessed with a fundus examination or retinal photography performed within 6 months before selection or before the randomisation at the latest) with visual impairment which could compromise the safety of rapid glucose control normalisation and the compliance to the study,
10. Planned initiation of a treatment that would impact the blood glucose levels (such as steroids) during the study period,
11. Patient deprived of liberty by a judicial or administrative decision, patient admitted to a social institution or who is under a measure of legal protection, patient hospitalized without consent or who is in an emergency situation.
12. Lack of effective contraception in women of childbearing potential,
13. Subject with a history of hearing or vision impairment hindering perception of glucose display and alarms (as this point is a contra-indication stated in the user's manual of the investigational medical device),
14. Severe impairment of renal function (Creatinine Clearance < 30 mL/min),
15. Patient on dialysis (as the user's manual of Dexcom G6 states that G6 readings may be inaccurate in this population)
16. Conditions which may increase the risk of induced hypoglycemia as per the investigator's judgment,
17. lnpatient psychiatric treatment in the past 6 months,
18. Current or recent abuse of alcohol or recreational drugs,
19. Patients that have frequent exposure to magnetic resonance imaging (MRl), computed tomography (CT) scan, or high frequency electrical heat (diathermy) treatment (as this point is a contra-indication stated in the user's manual of the investigational medical device and Dexcom G6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves REZNIK, Pr, Principal Investigator — CHU CAEN
Locations (10):
- France (10):
  - CHRU Brest, Brest, Brittany Region
  - CHU Rouen, Rouen, Normandy
  - CHU Amiens, Amiens, Picardie
  - CHU Caen, Caen
  - Hopital Européen de Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Nancy-Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - APHP Lariboisière, Paris, Île-de-France Region

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 patients were enrolled from 8 centres in one country (France). Among them, 30 patients were randomized, 15 in each study group. Following randomization in the experimental intervention group, one patient withdrew consent before insulin pump installation and effective start of study follow-up.
  First Patient Enrolled: December 30, 2019 - Last Patient Completed: May 30, 2022
Groups:
- Closed-loop and Home Care Services: automated insulin delivery system (Closed-loop) with tailored Home Healthcare Provider (HHP) services
  t:slim X2 with Control-IQ: closed-loop in patients at home for three months
  home healthcare services: home healthcare services from Air Liquide subsidiaries in patients at home for three months
Period: Overall Study
Arm/Group | Usual Care | Closed-loop and Home Care Services
Started | 15 | 14
Completed | 14 | 11
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Exclusion criterion found the day after initiation visit | 1 | 0
Not completed — Lack of complance to study procedures and less than 14 days on closed-loop | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Closed-loop and Home Care Services | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.3) | 69.3 (6.7) | 69.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 2 | 7 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 15 | 14 | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.62 (6.51) | 32.26 (4.33) | 34.00 (5.73)
HbA1c [Mean (Standard Deviation); unit: percentage of blood glycated haemoglobin] | 9.25 (1.04) | 8.98 (1.17) | 9.12 (1.09)
Time since Type 2 Diabetes diagnosis [Mean (Standard Deviation); unit: years] — Time between the date of Type 2 Diabetes diagnosis and the date of study selection visit expressed in years
  years | 16.97 (9.05) | 20.39 (12.28) | 18.62 (10.67)
Time since insulin therapy onset [Mean (Standard Deviation); unit: years] — Time between the date of insulin therapy first prescription and the date of study selection visit expressed in years
  years | 9.39 (8.03) | 8.99 (10.19) | 9.20 (8.97)
Number of daily insulin injections, basal [Mean (Standard Deviation); unit: number of injections] | 1.0 (0.0) | 1.1 (0.4) | 1.1 (0.3)
Number of daily insulin injections, bolus [Mean (Standard Deviation); unit: number of injections] — Population: In the experimental intervention group, 12 patients out of 14 were on concomitant insulin bolus scheme.
  number of injections
    number analyzed (Participants) | 15 | 12 | 27
    (all) | 2.7 (0.6) | 2.9 (0.3) | 2.8 (0.5)
Patient previously using continuous glucose monitoring [Count of Participants; unit: Participants] | 8 | 5 | 13
Patient with at least one concomitant blood glucose lowering drug [Count of Participants; unit: Participants] | 12 | 8 | 20
Patient on metformin [Count of Participants; unit: Participants] | 9 | 6 | 15
Patient on glucagon-like peptide-1 analogues [Count of Participants; unit: Participants] | 6 | 4 | 10
Patient on concomitant treatment for cardiovascular disease [Count of Participants; unit: Participants] | 14 | 14 | 28
Patient with at least one cardiovascular comorbidity [Count of Participants; unit: Participants] | 12 | 13 | 25
Patient with at least one concomitant cardiac disorder [Count of Participants; unit: Participants] | 5 | 5 | 10
Patient with at least one diabetes-related comorbidity [Count of Participants; unit: Participants] | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Time in Range (TIR)
Description: Time In Range, defined as the percentage of time spent with glucose measurements at 70-180 mg/dL (3.9-10.0 mmol/L) recorded by continuous glucose monitoring (CGM), during the last 14 days completed CGM recording from days 70 to 90
Time Frame: From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time | 36.61 (21.99) | 63.03 (9.41)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and Time In Range (TIR) at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p < .001, ANCOVA — Study group effect; Adjusted means difference = 27.4, 95% CI 2-sided [15.0 to 39.8], Standard Error of Mean 6.0 — Between-group adjusted means difference is calculated as analysis of covariance adjusted mean in Intervention Group - adjusted mean in Usual Care Group

2. Secondary Outcome: Time in Range (TIR) During Diurnal Period
Description: Time in range during diurnal period (06.00-23.59), defined as the percentage of time spent with glucose measurements at 70-180 mg/dL (3.9-10.0 mmol/L) recorded by continuous glucose monitoring (CGM), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 37.48 (23.46) | 34.30 (21.60)
  From days 70 to 90 | 36.96 (20.57) | 60.19 (10.96)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and Time In Range (TIR) during diurnal period at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p < .001, ANCOVA — Study group effect; Adjusted means difference = 23.0, 95% CI 2-sided [10.6 to 35.5], Standard Error of Mean 6.0 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time in Range (TIR) During Nocturnal Period
Description: Time in range during nocturnal period (00.00-05.59), defined as the percentage of time spent with glucose measurements at 70-180 mg/dL (3.9-10.0 mmol/L) recorded by continuous glucose monitoring (CGM), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 43.20 (31.23) | 34.82 (25.24)
  From days 70 to 90 | 35.56 (30.18) | 71.56 (15.04)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and Time In Range (TIR) during nocturnal period at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p < .001, ANCOVA — Study group effect; Adjusted means difference = 40.8, 95% CI 2-sided [25.8 to 55.8], Standard Error of Mean 7.2 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time Above Range (TAR) (Above 180 mg/dL)
Description: Time above target range defined as the percentage of time spent with CGM glucose measurements >180 mg/dL (10.0 mmol/L), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 60.43 (23.73) | 64.59 (21.54)
  From days 70 to 90 | 62.69 (22.91) | 36.14 (8.52)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and Time Above Range (TAR) at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p < .001, ANCOVA — Study group effect; Adjusted means difference = -27.7, 95% CI 2-sided [-40.5 to -15.0], Standard Error of Mean 6.1 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time Above Range (TAR) (Above 250 mg/dL)
Description: Time above target range defined as the percentage of time spent with CGM glucose measurements ≥250 mg/dL (13.9 mmol/L), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 30.21 (28.35) | 31.76 (23.37)
  From days 70 to 90 | 28.50 (22.35) | 9.12 (6.13)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.003, ANCOVA — Study group effect; Adjusted means difference = -20.1, 95% CI 2-sided [-32.4 to -7.9], Standard Error of Mean 5.9 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time Below Range (TBR) (Below 70 mg/dL)
Description: Time below target range, defined as the percentage of time spent with CGM glucose measurements <70 mg/dL (3.9 mmol/L), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 0.65 (1.08) | 0.98 (1.64)
  From days 70 to 90 | 0.70 (1.27) | 0.83 (1.47)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and Time Below Range (TBR) at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p = 0.79, ANCOVA — Study group effect; Adjusted means difference = 0.1, 95% CI 2-sided [-1.0 to 1.3], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time Below Range (TBR) (Below 54 mg/dL)
Description: Time below target range, defined as the percentage of time spent with CGM glucose measurements <54 mg/dL (3.0 mmol/L), during the last 14 days completed CGM recording at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of time
  At baseline | 0.14 (0.29) | 0.59 (1.59)
  From days 70 to 90 | 0.17 (0.42) | 0.18 (0.46)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.84, ANCOVA — Study group effect; Adjusted means difference = 0.0, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.2 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Glucose Variability (% CV Coefficient of Variation)
Description: Glucose variability assessed by coefficient of glucose variation (% CV) calculated by dividing the Standard Deviation (SD) by the corresponding mean of the CGM glucose measurements during the last 14 days at the end of the selection period (baseline before randomisation) and the last 14 days from days 70 to 90
Time Frame: At baseline and From days 70 to 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of coefficient of variation
  At baseline | 28.22 (7.34) | 29.45 (5.00)
  From days 70 to 90 | 28.22 (3.86) | 31.51 (5.69)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and glucose variability (% CV Coefficient of Variation) at baseline (during the last 14 days completed continuous glucose monitor recording at the end of the study selection period); p = 0.060, ANCOVA — Study group effect; Adjusted means difference = 3.7, 95% CI 2-sided [-0.2 to 7.6], Standard Error of Mean 1.9 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: HbA1c
Description: Blood glycated Haemoglobin A1c (HbA1c) value assayed in % at initiation visit (day 0) and at day 90
Time Frame: On day 0 and day 90
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
percentage of glycated haemoglobin
  On day 0 | 9.16 (1.01) | 9.03 (1.31)
  On day 90 | 8.79 (1.01) | 7.42 (0.64)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model with 2 factors: HbA1c value at baseline and study group; p < .001, ANCOVA — Study group effect; Adjusted means difference = -1.3, 95% CI 2-sided [-1.9 to -0.7], Standard Error of Mean 0.3 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Total Daily Insulin Dose
Description: Total daily insulin dose (expressed in IU/day) calculated as the sum of daily dose of insulin injections recorded by investigators whether basal, bolus or premix at selection (baseline) and study end (planned on day 90) visits
Time Frame: At selection (baseline) and study end (day 90) visits
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: IU/day
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
IU/day
  At selection visit: number analyzed (Participants) | 12 | 11
  At selection visit | 80.3 (39.5) | 66.8 (39.2)
  At study end visit | 111.7 (72.4) | 80.6 (61.8)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and total daily insulin dose at selection; p = 0.52, ANCOVA — Study group effect; Adjusted means difference = -18.5, 95% CI 2-sided [-78.2 to 41.2], Standard Error of Mean 28.5 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Body Weight
Description: Body weight (expressed in kg) recorded by investigators at initiation (day 0) and study end (planned on day 90) visits
Time Frame: At initiation (day 0) and study end (day 90) visits
Population: Efficacy intention to treat data set: all randomized patients followed-up at least 2 weeks after their randomization
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Closed-loop and Home Care Services
Number analyzed (Participants) | 14 | 11
kg
  At initiation visit | 92.10 (17.29) | 86.05 (20.87)
  At study end visit | 91.34 (17.81) | 87.66 (21.07)
Statistical Analysis 1: Comparison: Usual Care vs Closed-loop and Home Care Services; Test type: Superiority — Analysis of covariance (ANCOVA) model adjusted on the HbA1c stratification factor and body weight at study initiation visit; p = 0.08, ANCOVA — Study group effect; Adjusted means difference = 2.8, 95% CI 2-sided [-0.4 to 6.1], Standard Error of Mean 1.6 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the signature of the informed consent to the study end (planned on day 90) for each participating patient
Arm/Group | Usual Care | Closed-loop and Home Care Services
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/15 | 5/14
Other Adverse Events (participants affected / at risk) | 7/15 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=15) | Closed-loop and Home Care Services (N=14)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=15) | Closed-loop and Home Care Services (N=14)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 4 (4)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Device connection issue (Product Issues) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the Sponsor can review results communications prior to public release. According to Article R.5121-13 of the French Public Health Code, the results of the Research may not be published or the subject of written or oral communications by the PI without prior written consent of the Sponsor. The disclosure restriction applies to the Parties during the entire duration of the agreement and as long as the confidential data are not in the public domain.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04233229/Prot_SAP_000.pdf